CLINICAL TRIAL: NCT01954225
Title: Role of Udumbara Sutra in the Management of Fistula in Ano a Rare Case Study
Acronym: Bhagandara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Ayurved College and Hospital (Other Government)
Responsible Party: Principal Investigator, Dr.Nita Mahadevrao Kedar, Associate professor, Government Ayurved College and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1314
Record Dates: First submitted 2013-09-06; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Fistula in Ano
Keywords: Fistula in ano; Bhagandara; Udumbara sutra
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Udumbara sutra (Other): The Udumbara Sutra is a standard medicated thread smeared with latex of Udumbara (Ficus Glomerata) which has cutting and healing property.
  Interventions: Other: Udumbara Sutra

INTERVENTIONS:
Other: Udumbara Sutra — The Udumbara sutra is a standard medicated thread smeared with latex of Udumbara (Ficus Glomerata) which has cutting and healing property.
  Other Names: Medicated Thread

SUMMARY:
The anal fistula is a notorious disease due to its recurrence rate. Bhagandara is varyingly defined as a tear, ulcer or boil at Bhaga (Perianal region) within 2 finger circumference of it, causing painful abscess when opened is called Bhagandara. The Sanskrit word 'Bhagandara' has got two components-Bhaga and Darana. Bhaga means perianal region and Darana means to tear. The ancient Surgeon Sushruta has advocated various types of operations in Sushruta Samhita. He has advocated Kshara Sutra treatment due to probability of recurrence after surgery. Sushruta describes many kind of kshara like Palasa, Kadali. The most remarkable is Udumbara( Ficus Glomerata) among them. The present treatment modality Udumbara Kshara Sutra has been found effective due to its action of proper drainage of pus from the fistula that leads to a proper healing and as adjuvant therapy by avoid recurrence in Fistula in ano.

Hypothesis; Present treatment modality Udumber Sutra will found to be useful in tne management of Fistula in ano.

DETAILED DESCRIPTION:
A 5 year male child, come with complaints of painful discharging boil at left side of perianal region and pain with surgical history of incision and drainage for gluteal abscess done before six month. On local examination Patient had discharging sinus at 8 o' clock position on right side of Perianal region. Before planning the treatment other aetiologies were ruled out.

Under short general anaesthesia diagnosis was confirmed by probing as Fistula in ano. Internal opening of Fistula was confirmed by injecting Methylene Blue dye through external opening. The track was directed upward in the anal canal without any tributary. Length of the tract was 3cm, suggestive of low anal fistula.

Then Udumbara Sutra was tied covering the entire underlying track for cutting and healing under all aseptic precaution. The patient was discharged on the next day of procedure. The Udumbara Sutra was changed skilfully by weekly. To promote healing and to reduce pain and inflammation oral antibiotics, anti-inflammatory medicine were also prescribed.

The total period of Udumbara Sutra treatment was 1,1/2 month. The track cut through and simultaneously healed. The patient was observed for a period of 6 month to check for recurrence.

The Sutra or Medicated seton was a standard medicated thread smeared with latex of Udumbara (Ficus Glomerata), which has quality of cutting and healing.

ELIGIBILITY:
Inclusion Criteria:

* Patient without any major illness. Fistula in ano without tributaries ano without complication.

Exclusion Criteria:

* Multiple fistula and associated ano rectal conditions.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-02; Primary Completion 2006-04 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Use of Udumbara sutra in the management of Fistula in ano. | 1&1/2 month
  The Udumbara Sutra has good potential in the management by cutting and healing of Fistula in ano because it's less alkaline nature

SECONDARY OUTCOMES:
Use of Udumbara Sutra in avoiding recurrence of Fistula in ano | 1year
  Use Udumbara Sutra is found to be very effective in avoiding recurrence. There is no recurrence after one year.

CONTACTS AND LOCATIONS:
Overall Officials: Nita M Kedar, M.S.(Ayu), Principal Investigator — Associate Professor
Locations (1):
- Anand Surgical Hospital, Amravati, Maharashtra, India